CLINICAL TRIAL: NCT02268162
Title: Prospective Multicenter Randomized Control Study on Diagnosis of Individuals With Pulmonary Nodules by Different Bronchoscopy Combination
Brief Title: Diagnosis of Individuals With Pulmonary Nodules by Different Bronchoscopy Combination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); China Meitan General Hospital (Other); Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: lungcancer diagnosis; 201402024 (Other Grant/Funding Number: Ministry of Health in China)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Lung Neoplasms; Early Diagnosis; Bronchoscopy
Keywords: Lung Neoplasms; Bronchoscopy; Virtual Bronchoscopic Navigation(VBN); Fluoroscopy; Endobronchial Ultrasonography with a Guide Sheath(EBUS-GS); Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Routine Bronchoscopy (No Intervention): Participants in the group will receive routine bronchoscopy.
- Routine Bronchoscopy with a guiding equipment (Experimental): Participants in the group will receive routine bronchoscopy combined with a guiding equipment. These guiding equipments include virtual bronchoscopic navigation(VBN), endobronchial ultrasonography with a guide sheath(EBUS-GS) and fluoroscopy.
  Interventions: Procedure: guiding equipments
- Routine Bronchoscopy with two or more guiding equipments (Experimental): Participants in the group will receive routine bronchoscopy combined with two or more guiding equipments. These guiding equipments include virtual bronchoscopic navigation(VBN), endobronchial ultrasonography with a guide sheath(EBUS-GS) and fluoroscopy.
  Interventions: Procedure: guiding equipments

INTERVENTIONS:
Procedure: guiding equipments — The guiding equipments including VBN, EBUS-GS and fluoroscopy guide a bronchoscope along the bronchial route to a peripheral pulmonary lesion.
  Arms: Routine Bronchoscopy with a guiding equipment; Routine Bronchoscopy with two or more guiding equipments

SUMMARY:
This study evaluates the value of different bronchoscopy combination for diagnosing peripheral pulmonary lesions suspected to be cancer. One-third of participants will receive routine bronchoscopy, while one-third of participants will receive bronchoscopy combined with a guiding equipment and the other one-third of participants will receive bronchoscopy combined with two or more guiding equipments. These guiding equipments include virtual bronchoscopic navigation(VBN), endobronchial ultrasonography with a guide sheath(EBUS-GS) and fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects are adults with solitary peripheral pulmonary lesions (mean diameter, ≤30mm and >8mm from axial CT images) suspected to be cancer but were not pathologically confirmed.

Exclusion Criteria:

* Patient has dysrhythmia or cardiovascular disease that poses a risk during exercise.
* Patient has uncontrollable hypertension (SBP > 180mmHg).
* Patient has severe organ dysfunction (shock, severe hepatic and renal dysfunction, massive hemorrhage of upper gastrointestine, diffuse intravascular coagulation(DIC) and massive hemoptysis,etc).
* Patient has blood coagulation disorders (PT>2 times the upper limit of normal(ULN) or Platelet(PLT)<50000/ul）.
* Patient has severe dyspnea.
* Patient is allergic to local anesthetic.
* Patient is unable to provide informed consent.
* Patient is not an appropriate candidate for of is unable to tolerate flexible bronchoscopy procedures.
* Patient has any disease or condition that interferes with completion of initial or follow-up assessments of the effectiveness endpoints.
* Patient has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.
* Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study, or is currently participating in another clinical study.
* Female patient of childbearing potential has a positive result from a pregnancy test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3228 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield for pulmonary peripheral lesions | 7 days
  The diagnostic yield for individuals with pulmonary peripheral lesions examined by bronchoscopy with or without guiding equipments

SECONDARY OUTCOMES:
length of operation time using bronchoscopy or bronchoscopy combination | 30 minutes
  The operation time using bronchoscopy or bronchoscopy combination to examine a participant
length of stay in hospital | 7 days
  length of stay in hospital for a participant
hospitalization costs | 7 days
  the hospitalization costs for a participant
Number of participants with adverse events or serious adverse events | 2 weeks
  Number of participants with any adverse events or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Faguang Jin, MD & PhD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Asano F, Shinagawa N, Ishida T, Shindoh J, Anzai M, Tsuzuku A, Oizumi S, Morita S. Virtual bronchoscopic navigation combined with ultrathin bronchoscopy. A randomized clinical trial. Am J Respir Crit Care Med. 2013 Aug 1;188(3):327-33. doi: 10.1164/rccm.201211-2104OC. PMID 23600452
- [Background] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456
- [Background] Shinohara S, Hanagiri T, Takenaka M, Chikaishi Y, Oka S, Shimokawa H, Nakagawa M, Uramoto H, So T, Aoki T, Tanaka F. Evaluation of undiagnosed solitary lung nodules according to the probability of malignancy in the American College of Chest Physicians (ACCP) evidence-based clinical practice guidelines. Radiol Oncol. 2014 Jan 22;48(1):50-5. doi: 10.2478/raon-2013-0064. eCollection 2014 Mar. PMID 24587779